CLINICAL TRIAL: NCT04427956
Title: Prospective Randomised Corneal Crosslinking Study
Brief Title: Corneal Crosslinking Treatment Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNR2015/373
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-07

CONDITIONS: Progressive Keratoconus
Keywords: corneal crosslinking
MeSH Terms: interventions — Iontophoresis

STUDY DESIGN:
Intervention Model Description: Prospective randomized interventional clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Isotonic riboflavin (Active Comparator): CXL (UVA 9mW/cm2) treatment using isotonic riboflavin
  Interventions: Procedure: Corneal crosslinking: CXL (UVA 9mW/cm2); Drug: Isotonic riboflavin
- Hypotonic riboflavin (Active Comparator): CXL (UVA 9mW/cm2) using hypotonic riboflavin
  Interventions: Procedure: Corneal crosslinking: CXL (UVA 9mW/cm2); Drug: Hypotonic riboflavin
- Iontophoresis (Active Comparator): Iontophoresis with Ricrolin with following CXL (UVA 9mW/cm2).
  Interventions: Procedure: Corneal crosslinking: CXL (UVA 9mW/cm2); Procedure: Iontophoresis

INTERVENTIONS:
Procedure: Corneal crosslinking: CXL (UVA 9mW/cm2) — CXL treatment with UVA-radiation (9mW/cm2) with a 10 minute irradiation protocol.
Drug: Isotonic riboflavin — CXL protocol with isotonic riboflavin
  Arms: Isotonic riboflavin
Drug: Hypotonic riboflavin — CXL protocol with hypotonic riboflavin
  Arms: Hypotonic riboflavin
Procedure: Iontophoresis — CXL protocol with iontophoresis and ricrolin
  Arms: Iontophoresis

SUMMARY:
Three different protocols for inducing corneal crosslinks in subjets with progressive keratoconus will be evaluated in this randomised clinical study.

DETAILED DESCRIPTION:
Riboflavin does not penetrate the intact corneal epithelium. Corneal cross linking (CXL) is typically performed using the so-called "Dresden protocol". The Dresden protocol states 30 minutes of UVA-radiation (3mW/cm2) but a 10 minute irradiation protocol (9mW/cm2) is frequently used. Both of the protocols involve mechanical removal of the epithelium over the central 8 mm of the corneal surface. The first days after treatment therefore involves some degree of pain, often intense, and the presence of a healing epithelial defect may be associated with development of infiltrates in the cornea. A number of approaches have been evaluated in order to promote riboflavin penetration through the intact epithelium, of which iontophoresis appears most promising. Keratoconic corneas are thin at the cone location and sometimes it is difficult to maintain the safety margin of 400 microns during corneal crosslinking. Instead of using isotonic standard riboflavin, a swelling effect of the cornea can be obtained by using hypotonic riboflavin. However, the latter has been indicated as less effective in the process of inducing cross links.

Eighty-one of 81 patients of various degrees of keratoconus will be randomised to one of the following groups: 1) CXL (UVA 9mW/cm2) using isotonic riboflavin, or 2) CXL (UVA 9mW/cm2) using hypotonic riboflavin or 3) Iontophoresis with Ricrolin with following CXL (UVA 9mW/cm2).

Hypothesis:

i) CXL with hypotonic riboflavin or CXL with Ricrolin administered by iontophoresis or CXL with isotonic riboflavin is non-inferior compared to standard CXL with isotonic riboflavin.

ii) The morphological structure post-CXL in the three different groups will be similar without any significant differences.

The iontophoresis-assisted treatment arm has been interrupted due to low efficacy in halting disease progression. The results have been published.

ELIGIBILITY:
Inclusion Criteria:

* Progress in keratoconic eye. We define progress as an increase in Kmax of 1.0 diopter in 1 year or 0.5 diopter in 6 months. This increase in Kmax will be accepted as progression if concomitant changes tomographic parameters.

Exclusion Criteria:

* Concurrent ocular infection or corneal disease other than keratoconus.
* Pregnancy.
* Treatment with Isotretinoin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Postoperative change in visual acuity | Patients will be evaluated 1, 6, 12 and 24 months after treatment.
  Uncorrected visual acuity (UCVA) and best spectacle corrected visual acuity (BSCVA)
Postoperative change in Kmax | Patients will be evaluated 1, 6, 12 and 24 months after treatment.
  Maximum corneal steepness

SECONDARY OUTCOMES:
Postoperative change in astigmatism | Patients will be evaluated 1, 6, 12 and 24 months after treatment.
  Corneal astigmatism
postoperative change in corneal nerve cell density | Confocal microscopy will be performed at 6 and 12 months.
  Corneal nerve cell density will be evaluated using confocal microscopy
Postoperative change in Keratocyte cell density | Confocal microscopy will be performed at 6 and 12 months.
  Keratocyte cell density will be evaluated using confocal microscopy
Postoperative change in endothelial cell count | Confocal microscopy will be performed at 6 and 12 months.
  Endothelial cell count will be evaluated using confocal microscopy
Postoperative change in demarcation lines | Confocal microscopy will be performed at 6 and 12 months.
  Identification of the demarcation lines with confocal microscopy will help establishing how deep was the effect of the CXL treatment.
Postoperative change in the corneal thickness during CXL treatment | Corneal pachymetry will be evaluated before and then every 5 minutes during 30 minutes under CXL treatment.
  Corneal pachymetry is the process of measuring the thickness of the cornea

CONTACTS AND LOCATIONS:
Overall Officials: Ingemar Gustafsson, MD, Principal Investigator — Region Skåne
Locations (1):
- Skåne University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gustafsson I, Ivarsen A, Hjortdal J. Early findings in a prospective randomised study on three cross-linking treatment protocols: interruption of the iontophoresis treatment protocol. BMJ Open Ophthalmol. 2023 Sep;8(1):e001406. doi: 10.1136/bmjophth-2023-001406. PMID 37739426